CLINICAL TRIAL: NCT05574530
Title: A Colon-delivered Multivitamin Supplement to Support Vigilance and Cognitive Performance Under Stressful Working Conditions in Military Subjects
Brief Title: Vitamin (VIT) for Vigilance Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University and Research (Other)
Collaborators: Radboud University Medical Center (Other); Dutch Ministry of Defense (Unknown); DSM (Unknown); Thales (Unknown); Circadian (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NL75954.091.20
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Change; Stress
Keywords: Colon-delivered multivitamin supplement; Cognitive performance; Vigilance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Supplements are labeled A and B by a scientist who is not involved in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colon-delivered multivitamin supplement (Experimental): Colon-delivered multivitamin mix with vitamin B2, B3, B6, B9, vitamin C and D3. These vitamins are delivered as capsules coated by a eudragit S100 coating layer, in order to prevent systemic absorption of the vitamins in the small intestine.
  Interventions: Dietary Supplement: Colon-delivered multivitamin supplement
- Placebo supplement (Placebo Comparator): Placebo supplement containing microcrystalline cellulose, coated in the same way as the experimental product in order to prevent systemic absorption in the small intestine.
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Colon-delivered multivitamin supplement — 6-week intervention of one dietary supplement a day, containing vitamin B2 (10mg), vitamin B3 (4mg), vitamin B6 (1.4mg), vitamin B9 (400μg), vitamin C (200mg) and vitamin D3 (15ug).
  Arms: Colon-delivered multivitamin supplement
Dietary Supplement: Placebo supplement — 6-week intervention of one dietary supplement a day, containing 200 mg of microcrystalline cellulose.
  Arms: Placebo supplement

SUMMARY:
This study aims to examine the effects of a 6-week colon-delivered multi-vitamin supplement intervention on cognitive performance and stress levels in military under real-life, stressful working conditions.

The study is a randomized, double-blind, placebo-controlled, parallel trial in a real-life setting (military field exercise). The intervention product is a nutritional supplement, composed of vitamins B2, B3, B6, B9, C, and D3. These vitamins will be delivered in the colon where most of these vitamins can be utilized by the gut microbiota, as they act as cofactors for important cellular functions.

The main study outcome is the backward digit span (DS) score in a cognitive test, during the field exercise as compared to the start of the 6-week supplementation period. Secondary parameters are other cognitive test scores and a combined (z-scored) cognitive performance score. Stress levels will be measured in salivary cortisol and self-perceived stress levels will be derived from the HADS and PSS-10 questionnaire. Other stress biomarkers (e.g. heart rate variability) will be measured by a wearable.

DETAILED DESCRIPTION:
A growing number of professionals work in a type of job that brings psychological or physical stress while requiring optimal alertness and cognitive control, so called vigilance. These professionals are for example found in military contexts. Even a tiny lapse in alertness can carry large risks for themselves and others. Some studies suggest that dietary supplementation interventions can support shifts in the gut microbiome composition, leading to beneficial effects on various aspects of cognitive performance.

The primary objective in this study is to examine the effects of a 6-week colon-delivered multi-vitamin supplement intervention on cognitive performance and stress levels in military under real-life, stressful working conditions. The hypothesis here is that increased delivery of the nutrients in the colon can support the microbe community and complement microbe metabolites production (e.g. Short Chain Fatty Acids) that via the gut-brain axis support cognitive performance. A secondary objective is to investigate whether 6-week supplementation of the colon-delivered multivitamin mix reduces stress levels during the field exercise and cognitive tests.

The study is a randomized, double-blind, placebo-controlled, parallel trial in a real-life setting (military field exercise). The intervention product is a nutritional supplement, composed of vitamins B2, B3, B6, B9, C, and D3. The main study outcome is the backward digit span (DS) score in a cognitive test, during the field exercise as compared to the start of the 6-week supplementation period. Secondary parameters are other cognitive test scores and a combined (z-scored) cognitive performance score. Stress levels will be measured in salivary cortisol and self-perceived stress levels will be derived from the HADS and PSS-10 questionnaire. Other stress biomarkers (e.g. heart rate variability) will be measured by a wearable.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-50 years old
* Participating in military field exercise
* BMI between 18.5 - 30 kg/m2
* Stable body weight (< 5 kg change) over the past 3-months;

Exclusion Criteria:

* Food allergies or other issues with foods that would preclude intake of the study products
* History of gastro-intestinal surgery or gastro-intestinal complaints or gastrointestinal diseases (i.e., diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers)
* Suffering from metabolic, neuro-psychiatric disease (i.e., diabetes, hepatitis, HIV, cancer, epilepsy, major depression, AD(H)D, schizophrenia, etc.)
* Taking medication related to gut diseases or stress
* Being severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
* Use of antibiotics within the previous 3 months
* Not willing to refrain from taking other supplements during the intervention period
* Pregnant, lactating or having a wish to become pregnant during the study
* History of drug and/or alcohol abuse at the time of enrolment
* Using doctor described drugs related to gut or neurological/psychiatric diseases
* Alcohol intake > 3 servings of alcoholic beverages per day
* Planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study
* Suffering from an eating disorder
* Vegetarian/vegan diet or other issues with foods that would preclude intake of the study products
* High fibre diet (i.e. >30 g) based on our fibre intake screening tool
* Receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in backward digit span (DS) score | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  The backward DS score is related to working memory capacity. The score will be obtained from the forward/backward digit span cognitive task.

SECONDARY OUTCOMES:
Change in forward digit span (DS) score | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  The backward DS score is related to working memory capacity. The score will be obtained from the forward/backward digit span cognitive task.
Change in attention-switching task score | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Measuring interference control and cognitive flexibility
Change in Go-NoGo task score | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  By measuring response inhibition and sustained attention/vigilance
Change in overall cognitive performance score | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Calculate z-score from all three cognitive tests
Change in stress level | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Measured in salivary cortisol
Change in self-perceived stress levels | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Derived from the HADS and PSS10 questionnaire scores
Change in dietary fibre intake | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Derived from fibre screening questionnaire
Change in sleep quality | Baseline (before supplementation (T0)), after 5 weeks (T1) and after a field exercise after 6 weeks (T2)
  Derived from the Pittsburgh Sleep Quality Index questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No